CLINICAL TRIAL: NCT05434767
Title: Evaluating the Feasibility and Effectiveness of Using a Smartphone Application During Rehabilitation in Patients After Total Knee Replacement: A Pilot Feasibility Randomized Controlled Trial
Brief Title: Evaluating the Feasibility and Effectiveness of Using a Smartphone Application During Rehabilitation in Patients After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/2718
Record Dates: First submitted 2022-06-15; First posted 2022-06-28 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Total Knee Replacement; Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rehabilitation program (Active Comparator)
  Interventions: Other: Standard rehabilitation program
- Mobile application (Experimental)
  Interventions: Device: Mobile application

INTERVENTIONS:
Device: Mobile application — Participants will be instructed on the installation and use of the mobile application on their personal mobile phones. Participants will then have to perform the assigned exercises using the mobile application 3 times daily. Physiotherapists will still perform the required assessment/review, education, and intervention.
  Arms: Mobile application
Other: Standard rehabilitation program — All participants will be seen by physiotherapists in the ward post-TKR surgery and undergo standard inpatient rehabilitation. Patients will be given instructions to perform assigned exercises 3 times daily. Physiotherapists will perform the required assessment/review, education, and intervention.
  Arms: Standard rehabilitation program

SUMMARY:
Despite best efforts to provide standardized and effective rehabilitation sessions post-total knee replacement (TKR), there are a few factors that may result in sub-optimal recovery in this group of patients. There is a need to develop innovative rehabilitation strategies that (i) provide patients with accurate cues allowing for better compliance and exercise performance, (ii) allow for therapists to ensure continuity of care, monitor compliance, and identify deviation from recovery trajectories post-discharge, prior to their first outpatient appointment, and (iii) reduce reliance on manpower and variability during rehabilitation sessions.

Technological solutions that empower patients and allow home-based rehabilitation to take place without the need for real-time human supervision could be the key to improving effectiveness and lowering costs. A mobile application which detects key landmarks on the body for human pose estimation will allow patients to perform their rehabilitation exercises with real-time feedback allowing for proper execution of the exercises. Physiotherapists will be able to access the data generated from the exercise session via a command centre to monitor patients' recovery progress and compliance.

The primary aim of this pilot study is to evaluate the feasibility of using a mobile application during rehabilitation in patients after a TKR surgery. The secondary aim is to study the effects of using a mobile application during rehabilitation on knee functional status, exercise self-efficacy, and treatment satisfaction after TKR surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Primary unilateral total knee replacement
2. Age >= 45 years
3. Under the Enhanced Recovery After Surgery (ERAS) programme (discharge on post-operative day 0/1)
4. Willingness to be randomized to either mobile application group or standard hospital-based rehabilitation group
5. Ability to provide informed consent
6. Is technologically savvy - at least 6 months' experience using a smartphone and able to key in data into a smartphone
7. English-speaking

Exclusion Criteria:

1. Rheumatoid arthritis and other systemic arthritis
2. A previous history of stroke and other major neurological conditions
3. An intention to transfer to step-down care facilities post-operatively or intention to continue outpatient physiotherapy service at another institution
4. Unable to perform 5 repetitions of inner-range quadriceps exercise

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Compliance | 6 weeks post-surgery
  Frequency of exercise sessions completed

SECONDARY OUTCOMES:
Knee range-of-motion | Pre-operation; 6 weeks post-surgery
  A long-arm goniometer will be used to measure knee flexion and extension range-of-motion.
Gait speed | Pre-operation; 6 weeks post-surgery
  Usual and fast gait speed
Knee Pain | Pre-operation; 6 weeks post-surgery
  Knee will be measured using separate 11-point numeric pain rating scale, with zero representing no pain at all and 10 representing worst imaginable pain.
30 second sit to stand | Pre-operation; 6 weeks post-surgery
  30 second sit to stand test
Self-report physical function | Pre-operation; 6 weeks post-surgery
  All items are scored on 5-point Likert scales. With100 indicating no symptoms and 0 indicating extreme symptoms.
Self-efficacy | Pre-operation; 6 weeks post-surgery
  Self-efficacy questionnaire
Total contact time | 6 weeks post-surgery
  Time spent with the patients
Quality of the mobile application | 6 weeks post-surgery
  Quality of the mobile application questionnaire. All items are scored on 5-point Likert scales with 1 indicating "Inadequate" and 5 indicating "Excellent".
Participant satisfaction | 6 weeks post-surgery
  Participants will rate their satisfaction with treatment on an 11-point Likert scale, with 0 indicating "no satisfaction" and 10 indicating "complete satisfaction".
Treatment credibility | 6 weeks post-surgery
  Participants will rate their confidence about the benefits of the intervention on an 11-point Likert scale, with 0 indicating "not confident" and 10 indicating "extremely confident".
Perceived usefulness and ease of use | 6 weeks post-surgery
  Participants will rate their perceived usefulness and ease of use of the intervention on an 11-point Likert scale, with 0 indicating "not useful or not easy" and 10 indicating "extremely useful or extremely easy".

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided